CLINICAL TRIAL: NCT00112177
Title: A Multicentre, Randomized, Double-Blind Placebo-Controlled Study of the Efficacy and Safety of Itopride HCl in Patients Suffering From Functional Dyspepsia
Brief Title: Effect of Itopride, on Symptoms of Functional Dyspepsia, Such as Indigestion, Bloating, Inability to Finish a Meal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Monique Giguère, Axcan Pharma inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITOFD04-03
Record Dates: First submitted 2005-05-31; First posted 2005-06-01 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Dyspepsia
Keywords: Functional dyspepsia; Abdominal Symptom relief; Fullness; Bloating; Indigestion
MeSH Terms: conditions — Dyspepsia | interventions — itopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Itopride Hydrochloride

SUMMARY:
Itopride is a new compound that is already marketed in Japan and in some countries of Eastern Europe under the name of Ganaton. It is used to treat symptoms of functional dyspepsia. Patients suffering from this condition have difficulties digesting food. They feel full after eating a few bites; they feel bloated and their stomachs hurt. The goal of this study is to see if itopride helps to relieve the symptoms of functional dyspepsia.

DETAILED DESCRIPTION:
The study lasts approximately 10 weeks. Patients may either receive the real itopride, or a sugar pill called placebo. They have equal chances of receiving either treatment. After having completed this study, patients may be eligible to continue treatment for a longer period. At that point, all patients receive itopride.

Patients need to come to the clinic for evaluations 4 times during the trial. Various evaluations are done at these visits, such as a physical exam, lab tests, evaluation of the heart condition, and questionnaires need to be completed by the patient to see if the drug helps them in relieving their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from functional dyspepsia according to Rome II criteria

  * 18-65 years old
  * Absence of, or infrequent heartburn (one episode per week or less)
  * Helicobacter pylori (H. pylori) negative
  * Normal upper endoscopy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Symptom relief

SECONDARY OUTCOMES:
Impact of symptom relief on quality of life
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Professor, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Monique Giguère, Ph.D. - Programs Director, Mont-Saint-Hilaire, Quebec, Canada